CLINICAL TRIAL: NCT04410302
Title: University of California Minority Patient-Derived Xenograft (PDX) Development and Trial Center (UCaMP) to Reduce Cancer Health Disparities
Brief Title: Patient-Derived Xenografts to Reduce Cancer Health Disparities
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of California, Davis (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1420270; NCI-2020-01323 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 1420270-1 (Other: University of California Davis Comprehensive Cancer Center); P30CA093373 (NIH); U54CA233306 (NIH)
Record Dates: First submitted 2020-05-27; First posted 2020-06-01 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: Bladder Carcinoma; Gastric Carcinoma; Liver and Intrahepatic Bile Duct Carcinoma; Lung Carcinoma; Malignant Neoplasm
MeSH Terms: conditions — Urinary Bladder Neoplasms; Stomach Neoplasms; Carcinoma, Hepatocellular; Lung Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Tumor tissue, blood, saliva, urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Ancillary-correlative (biospecimen collection): Patients undergo collection of tumor tissue samples during standard of care tumor biopsy or surgical resection to establish PDXs. Patients may also undergo collection of blood, saliva, and urine samples to compare DNA abnormalities to noncancer cells in order to determine if they were present before the cancer started or developed with it.
  Interventions: Procedure: Biospecimen Collection

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of tumor tissue, blood, saliva, and urine samples

SUMMARY:
This trial establishes patient-derived cancer xenografts in addressing cancer health and treatment disparities that disproportionately affect racial/ethnic minorities. Understanding the genetic and response differences among racial/ethnic minorities may help researchers enhance the precision of therapeutic treatments.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Develop and characterize over 200 patient-derived xenografts (PDXs), with at least 50 PDXs each for gastric, liver, bladder, and lung cancers with 60% (approximately) of the PDXs from minority patients, focusing on Hispanic/Latino Americans [HLAs], African Americans [AAs], and Asian American/Native Hawaiians/Pacific Islanders [AANHPIs].

II. Utilize these PDXs in preclinical testing of single agents and drug combinations to guide precision cancer medicine decision-making with a focus upon the predominant racial/ethnic minority populations residing in California compared to non-Hispanic Whites [NHWs].

III. Conduct "Characterizing Treatment Responses with PDX Models for Gastric and Liver Tumors" as Research Project 1, focused on the most common histological forms of gastric cancer (GC) and liver cancers (LC) primarily from HLAs and AANHPI patients.

IV. Conduct "Characterizing Treatment Responses with PDX Models for Lung and Bladder Tumors" as Research Project 2, focused on lung squamous cell carcinoma (LSCC) and advanced urothelial or bladder cancer (aBC) primarily from AA and NHW patients.

V. Collaborate with the National Cancer Institute (NCI), other PDX Development and Trial Centers (PDTCs), non-PDXNet, PDXNet Data Commons and Coordinating Centers to fulfill the mission of the PDXNet.

VI. Select and conduct pilot projects through the Pilot Projects and Trans-Network Activities Core (PPTNAC) inclusive of UCaMP members, other PDTCs and beyond that will evaluate comparative therapeutic responses using PDX models and contribute to the elucidation of biological determinants of cancer health disparities in gastric, liver, bladder, and lung cancers.

OUTLINE:

Patients undergo collection of tumor tissue samples during standard of care tumor biopsy or surgical resection to establish PDXs. Patients may also undergo collection of blood, saliva, and urine samples to compare deoxyribonucleic acid (DNA) abnormalities to noncancer cells in order to determine if they were present before the cancer started or developed with it.

ELIGIBILITY:
Inclusion Criteria:

* Patient receiving treatment for the above 4 cancers (bladder cancer, lung cancer, gastric/stomach cancer, and liver cancer)
* Signed informed consent that will be put on file

Exclusion Criteria:

* No informed consent obtained
* Specimen unacceptable/degraded/etc.
* Individuals who are not yet adults (infants, children, teenagers)
* Pregnant women
* Prisoners
* Adults unable to consent

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with bladder cancer, lung cancer, gastric/stomach cancer, or liver cancer seen in routine clinic appointments within the University of California (UC) Davis Health System and contributing University of California Minority PDX (UCaMP) institutions
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-11-12 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Establish and characterize at least 200 patient-derived cancer xenografts (PDXs) | Up to 4 years
  The investigators will establish and characterize at least 200 PDXs, and utilize these PDXs in preclinicial testing of single agents and drug combinations that help guide future clinical decision-making emphasizing the largest racial/ethnic minority populations residing in California: Hispanic/Latino Americans ([HLAs), Asian Americans/Native Hawaiians/Pacific Islanders (AANHIPIs), and African Americans (AAs) compared to Non-Hispanic Whites (NHWs).

CONTACTS AND LOCATIONS:
Overall Officials: Luis G Carvajal-Carmona, Principal Investigator — University of California, Davis
Locations (2):
- United States (2):
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California